CLINICAL TRIAL: NCT06187961
Title: A Phase 2, Open-label, Single Arm Study of Combined HAIC, Lenvatinib and Cadonilimab As Conversion Therapy for Unresectable Hepatocellular Carcinoma
Brief Title: Combined HAIC, Lenvatinib and Cadonilimab As Conversion Therapy for Unresectable Hepatocellular Carcinoma
Acronym: CCGLC-011
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Akesobio (Industry)
Responsible Party: Principal Investigator, Ze-yang Ding, MD, Prof., Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-S039
Record Dates: First submitted 2023-12-08; First posted 2024-01-03 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Cadonilimab; Lenvatinib; Downstaging conversion therapy; Hepatocellular Carcinoma; Hepatic Arterial Infusion Chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAIC-len-cado (Experimental): Patients with advanced hepatocellular carcinoma who was initially evaluated unsuitable for the radical therapy and received combined HAIC plus lenvatinib (Len) and cadonilimab as conversion therapy for downstaging.
  Interventions: Procedure: HAIC; Drug: Lenvatinib plus cadonilimab

INTERVENTIONS:
Procedure: HAIC — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 3 weeks.
  Other Names: hepatic arterial infusion chemotherapy of FOLFOX
Drug: Lenvatinib plus cadonilimab — lenvatinib (8mg, qd) plus cadonilimab (10mg/kg, q3w)
  Other Names: levima plus cadonilimab

SUMMARY:
This is an open-label, single-arm, phase 2 study. The purpose of study is to evaluate the feasibility and safety of hepatic arterial infusion chemotherapy combined with lenvatinib and cadonilimab as conversion therapy for unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Cadonilimab is the world's first PD-1/CTLA-4 bispecific antibody tumor immunotherapy new drug, a tetrameric PD-1/CTLA-4 bispecific antibody, which can only bind to TIL tetravalent co-expressing PD-1 and CTLA-4. This design not only retains the efficacy observed in the combination therapy of PD-1 plus CTLA-4 inhibitors, but also reduces the risk of activated T cells attacking healthy tissues, thereby alleviating the toxicity problem outside the tumor. On June 29, 2022, the National Medical Products Administration of China approved the new drug Cadonilimab for the treatment of recurrent or metastatic cervical cancer patients who have failed platinum-based chemotherapy. Currently, a phase II clinical study of lenvatinib combined with Cadonilimab systemic treatment for advanced hepatocellular carcinoma is underway, and preliminary results reveal that in 30 enrolled patients, the ORR was 44.4%, the DCR was 77.8%, the treatment-related adverse reaction rate was 83.3%, but the incidence of grade 3 or above adverse reactions was only 26.7%. The safety of this antibody in patients is generally good. This study intends to evaluate the safety and efficacy of HAIC combined with lenvatinib and cadonilimab as a conversion regimen in unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma is proven on biopsy or confirmed by the presence of radiological hallmarks, according to the American Association for the Study of Liver Diseases or European Association for the Study of the Liver guidelines.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Not suitable for radical surgery (including radical hepatic resection, liver transplantation or liver cancer ablation) after evaluation by the hepatobiliary tumor MDT expert group. Specifically, any of the following conditions are met:

  1. R0 resection is not feasible.
  2. In subjects without cirrhosis, the volume of normal liver parenchyma is less than 30% of the total volume, or in subjects with cirrhosis, the volume of normal liver parenchyma is less than 40% of the total volume, or ICG-R15>15%.
  3. BCLC stage B or C: ①Multinodular HCC with Well defined nodules, preserved portal flow, selective access; ②Diffuse, infiltrative, extensive bilobar liver involvement; ③Portal invasion; ④>3 nodules or ≤3 nodules with at least one nodule>3cm.
* No prior systemic anti-tumor treatment for hepatocellular carcinoma before the first dose.
* According to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST V1.1), at least 1 measurable lesion, or a measurable lesion that has clearly progressed (based on RECIST V1.1 criteria) after local treatment.
* Subjects with portal vein tumor thrombus (PVTT):

  1. Chen's group A and B, or Cheng's type I-III can be enrolled.
  2. Chen's group C, or Cheng's type IV (superior vena cava tumor thrombus) cannot be enrolled.
* Subjects with hepatic vein tumor thrombus:

  1. VV1 and VV2 types can be enrolled.
  2. VV3 type, or Sakamoto type I (inferior vena cava tumor thrombus) can also be enrolled.
  3. Sakamoto type II (inferior vena cava tumor thrombus extending above the diaphragm), or Sakamoto type III (inferior vena cava tumor thrombus reaching the right atrium) cannot be enrolled.
* Subjects with oligometastases outside the liver can be enrolled: Oligometastases outside the liver are defined as up to three metastatic lesions in a maximum of two organs, with the largest diameter being 3cm.
* Child-Pugh score less than or equal to 7.
* Adequate organ and bone marrow function, with laboratory test values meeting the following requirements within 7 days prior to inclusion (no blood components, cell growth factors, albumin, or other intravenous or subcutaneous corrective treatment drugs are allowed within 14 days prior to obtaining laboratory tests):

  1. Complete blood count: Absolute Neutrophil Count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥75×10^9/L; Hemoglobin (HGB) ≥9.0 g/dL.
  2. Liver function: Total Bilirubin (TBIL) ≤2×Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤5×ULN; Serum albumin ≥28 g/L; Alkaline Phosphatase (ALP) ≤5×ULN.
  3. Kidney function: Serum Creatinine (Cr) ≤ 1.5×ULN or Clearance of Creatinine (CCr) ≥50mL/min (Cockcroft-Gault formula); Urinalysis shows proteinuria <2+; For subjects with baseline urinalysis showing proteinuria ≥2+, a 24-hour urine collection should be performed and 24-hour urinary protein quantification <1g.
  4. Coagulation function: International Normalized Ratio (INR) ≤2.3 or Prothrombin Time (PT) extension ≤6 seconds.
* Estimated life expectancy of ≥12 weeks.
* Female subjects of childbearing age or male subjects whose sexual partners are of childbearing age need to take effective contraceptive measures during the entire treatment period and for 6 months after the last medication.
* Signed written informed consent, and able to comply with the visit and related procedures stipulated in the protocol.

Exclusion Criteria:

* Histologically/cytologically confirmed fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc.
* History of hepatic encephalopathy or liver transplantation.
* Clinically symptomatic pleural effusion, ascites, or pericardial effusion requiring drainage. Subjects with only radiologically detected minimal pleural effusion, ascites, or pericardial effusion without symptoms can be enrolled.
* Acute or chronic active hepatitis B or C infection, with hepatitis B virus (HBV) DNA >2000IU/ml or 10^4 copies/ml; hepatitis C virus (HCV) RNA >10^3 copies/ml; co-positive for hepatitis B surface antigen (HbsAg) and anti-HCV antibody. Subjects who meet the above criteria after antiviral treatment with nucleoside analogs can be enrolled.
* Presence of central nervous system metastases.
* History of esophageal or gastric variceal bleeding due to portal hypertension within the past 6 months. Subjects assessed by the investigator to be at high risk of bleeding.
* Any life-threatening bleeding event within the past 3 months, including those requiring blood transfusion, surgery or local treatment, or continuous drug treatment.
* History of arterial or venous thromboembolic events within the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other serious thromboembolic events. Exceptions are made for thrombosis formation related to implanted venous infusion ports or catheters, or superficial vein thrombosis that has stabilized after routine anticoagulation treatment. Preventive use of low-dose low molecular weight heparin (such as enoxaparin 40 mg/day) is allowed.
* Continuous use of aspirin (>325 mg/day) or other known platelet function inhibitors such as clopidogrel or ticlopidine for 10 days within 2 weeks prior to the first dose.
* Uncontrolled hypertension, with systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
* Presence of any toxicity caused by previous treatment that has not recovered to grade 0 or 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE 5.0) before the first dose of study treatment (excluding alopecia, non-clinically significant and asymptomatic laboratory abnormalities).
* Symptomatic congestive heart failure (New York Heart Association class II-IV), left ventricular ejection fraction (LVEF) <50% as indicated by echocardiography.
* Symptomatic or poorly controlled arrhythmia. History of congenital long QT syndrome or corrected QTc >500 ms (calculated using the Fridericia formula) at screening.
* Severe bleeding tendency or coagulation disorder, or currently receiving thrombolytic therapy.
* History of gastrointestinal perforation and/or fistula, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive intestinal resection (partial colectomy or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within the past 6 months.
* Received radiotherapy within 3 weeks prior to the first dose of study treatment. For patients who received radiotherapy more than 3 weeks prior to the first dose of study treatment, all of the following conditions must be met for inclusion: no current radiation-related toxicities, no need for corticosteroids, and exclusion of radiation pneumonitis, radiation hepatitis, radiation enteritis, etc.
* History or current diagnosis of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of lung function, and other lung diseases.
* Active pulmonary tuberculosis, currently receiving anti-tuberculosis treatment, or received anti-tuberculosis treatment within 1 year prior to the first dose.
* Infection with human immunodeficiency virus (HIV) (HIV 1/2 antibody positive), known syphilis infection requiring treatment.
* Active or clinically uncontrolled severe infection. Severe infection within 4 weeks prior to the first dose, including but not limited to hospitalization for complications of infection, sepsis, or severe pneumonia.
* Active autoimmune disease requiring systemic treatment (such as disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) is allowed. History of primary immunodeficiency. Patients with only autoantibody positivity need to be confirmed by the investigator whether there is an autoimmune disease.
* Use of immunosuppressive drugs within 4 weeks prior to the first dose, excluding intranasal, inhaled, or other local corticosteroids or physiological doses of systemic corticosteroids (i.e., no more than 10mg/day prednisone or equivalent doses of other corticosteroids). Temporary use of corticosteroids for the treatment of dyspnea symptoms due to allergies or diseases such as asthma, chronic obstructive pulmonary disease, etc., is allowed.
* Received a live attenuated vaccine within 4 weeks prior to the first dose or planned to receive one during the study period.
* Major surgery (craniotomy, thoracotomy, or laparotomy) or unhealed wound, ulcer, or fracture within 4 weeks prior to the first dose. Minor surgical procedures or tissue biopsy within 7 days prior to the first dose, excluding venous puncture for the purpose of intravenous infusion, are excluded.
* Local treatment for hepatocellular carcinoma within 4 weeks prior to the first dose.
* Use of traditional Chinese medicine with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, etc., except for local use to control pleural effusion or ascites, etc.) within 2 weeks prior to the first dose.
* Other acute or chronic diseases, mental illnesses, or laboratory test abnormalities that may result in increased medical risk and/or uncertainty in survival assessment, or other conditions deemed by the investigator to be unsuitable for inclusion in the study.
* Diagnosis of other malignant tumors within 5 years prior to the first dose, excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or in situ carcinoma that has been radically resected. If other malignant tumors were diagnosed more than 5 years prior to the first dose, even if the liver lesions meet the clinical diagnostic criteria for hepatocellular carcinoma of the American Association for the Study of Liver Diseases (AASLD), pathological or cytological diagnosis of the liver lesions must be confirmed to be hepatocellular carcinoma for inclusion.
* Previous treatment with any anti-PD-1 antibody, anti-PD-L1/L2 antibody, anti-CTLA-4 antibody, or other immunotherapy. Previous treatment with targeted therapy against VEGF and/or VEGFR, RAF, MEK, PDGFR, FGFR, etc.
* Known allergy to any component of oxaliplatin, 5-fluorouracil, calcium folinate, lenvatinib, or cadonilimab; or severe allergic reaction to other monoclonal antibodies in the past.
* Patients diagnosed with aortic dissection aneurysm, celiac trunk and superior mesenteric artery dissection aneurysm.
* Received treatment in other clinical trials within 4 weeks prior to the first dose.
* Pregnant or breastfeeding women.
* Patients with systemic multiple metastases, portal vein tumor thrombus involving the superior mesenteric vein, inferior vena cava tumor thrombus extending above the diaphragm or reaching the right atrium.
* Other acute or chronic diseases, mental illnesses, or laboratory test abnormalities that may result in the following outcomes: increased risk associated with study participation or study drug administration, or interference with the interpretation of study results, and other conditions that make the patient ineligible to participate in the study based on the judgement of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Amendable to Curative Surgical Interventions | from the date of first treatment to the date of last treatment, an average of 3 years
  Number of patients amendable to curative surgical interventions defined as number of patients receiving curative surgical resection, transplantation, or ablation after successful down-sizing of tumor(s) by intervention.

SECONDARY OUTCOMES:
overall response rate (ORR) measured by mRECIST criteria | from the date of first treatment to radiographically documented progression according to mRECIST, assessed up to 3 years
  Complete response (CR): Disappearance of any intra-tumoral arterial enhancement in all target lesions; Partial response (PR): At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions; Stable disease (SD): Any cases that do not qualify for either partial response or progressive disease; Progressive disease (PD): An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started.
  ORR=CR+PR.
Overall survival (OS) | from the date of first treatment to the date of death from any cause, assessed up to 5 years
  Overall survival (OS): measured from date of first treatment to the date of death from any cause. Participants alive or lost to follow-up will be censored at the date of their last visit.
Progression-free survival (PFS) | from the date of first treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause, whichever occurs first, assessed up to 3 years
  measured from the date of first treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.
Time to progression (TTP) | from the date of first treatment to radiographically documented progression according to mRECIST, assessed up to 3 years
  Time to progression (TTP): measured from the date of first treatment to radiographically documented progression according to mRECIST 1.1. This does not include death from any cause.
Time to intrahepatic tumor progression (TTITP) | from the date of first treatment to radiographically documented intrahepatic tumor progression according to mRECIST, assessed up to 3 years
  Time to intrahepatic tumor progression (TTITP): measured from the date of first treatment to radiographically documented intrahepatic tumor progression according to mRECIST 1.1. This does not include death from any cause.
Incidence of Study-Related Adverse Events | from the date of first treatment to 90 days after last treatment, around 3 years and 90 days
  Incidence, nature, and severity of adverse events graded according to the United States National Cancer Institute The Common Terminology Criteria for Adverse Events (NCI-CTCAE 5.0)
Pathological complete response (pCR) | from the date of first study treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause, whichever occurs first, assessed up to 5 years
  Pathological response is assessed as the percentage of surface with non-viable cancer cells (represented by necrosis or fibrosis, the ultimate stage of necrosis) in relation to the total tumor area and will be equal to: 100% - viable cancer cells (%). If there are multiple tumors, the mean percentage will be used.
Disease control rate (DCR) | from the date of first treatment to radiographically documented response according to mRECIST, assessed up to 3 years
  Percentage of patients that had a CR, PR, or SD ≥ 6 months per mRECIST
Duration of response (DoR) | from the date of first documented evidence of CR or PR to first documented sign of PD or death from any cause according to mRECIST 1.1, assessed up to 3 years
  Defined as the time from first documented evidence of CR or PR until the first documented sign of disease progression (PD) or death from any cause
Quality of Life (QoL) after treatment | assessed form the date of first followup to radiographically documented progression or or death from any cause, up to 3 years
  The life quality of every subject is assessed every 3 months during follow up according to the 45-item FACT-Hep questionnaire, which assesses generic HRQL concerns and disease-specific issues.

CONTACTS AND LOCATIONS:
Overall Officials: Ze-yang Ding, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No